CLINICAL TRIAL: NCT03636282
Title: Hockey Fans in Training (Hockey FIT): A Pragmatic Cluster Randomized Controlled Trial to Improve Men's Health Through the Power of Sport
Brief Title: Hockey Fans in Training (Hockey FIT): Improving Men's Health Through the Power of Sport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Robert Petrella, Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 111881
Record Dates: First submitted 2018-07-25; First posted 2018-08-17 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Overweight; Obesity
Keywords: Chronic disease; Men's health; Health promotion; Exercise; Healthy diet; Health Technology; Weight loss; Hockey
MeSH Terms: conditions — Overweight; Obesity; Chronic Disease; Motor Activity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Pragmatic cluster randomized controlled trial with 2 arms: intervention (immediate delivery of Hockey FIT program) and comparator (wait-list control/delayed delivery of Hockey FIT program)
Who Masked: Outcomes Assessor
Masking Description: Trained assessors conducting measurements are not blinded to study allocation in all instances. When a trained assessor is not blinded, potential bias related to measurement of the primary outcome (weight) is being addressed by the requirement of photos of weight (measured via an electronic scale) being taken alongside the study measurement form (including study ID), at all follow-up time points. Furthermore, a study team member will verify that all weights recorded on the study measurement form match what is shown in the photo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hockey FIT Program (Immediate Delivery) (Experimental): Hockey FIT Program: A gender-sensitized, weight loss and healthy lifestyle program that engages men using the power of being a sports fan.
  Interventions: Behavioral: Hockey FIT Program (Immediate Delivery)
- Wait-List Control (Delayed Delivery) (No Intervention): No intervention for 12 months. After 12 months, Hockey FIT program is offered.

INTERVENTIONS:
Behavioral: Hockey FIT Program (Immediate Delivery) — Hockey FIT is comprised of a 3-Month Active Phase and a 9-Month Minimally-Supported Phase.
  Active Phase: 12 weekly, 90-minute group-based sessions consisting of classroom-based education and exercise. Outside of sessions, participants follow their individualized lifestyle prescriptions for healthy eating, physical activity (steps), and exercise. Participants are encouraged to regularly use health technology support tools customized to Hockey FIT. Minimally-supported phase: Participants are encouraged to continue with their healthy lifestyle behaviour changes and to regularly use the health technology support tools.
  Arms: Hockey FIT Program (Immediate Delivery)

SUMMARY:
Hockey Fans in Training (Hockey FIT) is a 12-month (3-month active phase and 9-month minimally-supported phase) weight loss and healthy lifestyle program for middle-aged, male hockey fans with overweight or obesity, delivered by trained coaches in collaboration with major junior or professional hockey teams and implementation partners (e.g., YMCAs, local fitness facilities, and universities) in Canada and the United States.

In the proposed study, a minimum of 32 sites (affiliated with hockey teams and local implementation partners) will be randomly assigned to either immediate delivery (Hockey FIT program) or delayed delivery (wait-list control). At each site, male hockey fans at risk for chronic diseases will be recruited to take part in the study (note: the goal is to recruit approximately 40 men/site). Sites assigned to the delayed delivery group will offer the Hockey FIT program to their enrolled participants after 12 months.

Through the Hockey FIT program, the investigators aim to promote weight loss, increase physical activity levels, and improve other health measures through a cost-effective solution that is acceptable and appealing to men who have overweight or obesity.

DETAILED DESCRIPTION:
The overall goal of this study is to reduce preventable chronic diseases in men by improving health behaviours and health indicators. To achieve this goal, following a successful pilot study providing strong evidence to proceed with a definitive trial, the investigators are conducting a pragmatic, cluster randomized controlled trial (RCT) of the Hockey FIT program.

The primary specific aim is to conduct an outcome evaluation to evaluate the effectiveness of Hockey FIT in middle-aged men who have overweight or obesity. Specifically, the investigators will: examine whether Hockey FIT (vs. wait-list control) leads to: greater weight loss at 12 months (primary outcome), as well as improved health behaviours (physical activity; sedentary time; eating habits) and health indicators (physiological measures; health & psychosocial measures) at 3 and 12 months.

Following the pilot study, the investigators will use the affiliation of being a fan of hockey as a powerful draw to engage men. Sites will be selected based on availability of both a major junior (or professional) hockey team and an implementation partner (e.g., YMCA branch, fitness facility, University) located in the city. A minimum of 32 sites in Canada and the United States will be randomized to the intervention (Hockey FIT program: immediately delivery) or comparator (wait-list control: delayed delivery); at each site, men will be recruited to participate (with the goal of recruiting approximately 40 men/site). Intervention sites will begin Hockey FIT immediately while comparator sites will offer Hockey FIT after a 12-month delay. The measurement sessions involving both groups will take place at 0 (baseline), 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male;
2. Between 35 and 65 years of age;
3. Objectively-measured body-mass index of at least 27 kg/m2
4. Deemed safe to participate in physical activity [i.e., clear the 2018 Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) or receive written clearance from a health care provider].

Exclusion Criteria:

1) Advised by a health care provider to not participate in the program

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 997 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Weight loss (absolute) | 12 months
  Measured using a digital weight scale (in kg)

SECONDARY OUTCOMES:
Weight loss (absolute) | 3 months
  Measured using a digital weight scale (in kg)
Weight loss (percent change) | 3 months & 12 months
  Measured using a digital weight scale (% change from baseline)
Predicted maximal oxygen uptake (VO2max) | 3 months & 12 months
  Calculated from sub-maximal fitness test (in mL/kg/min)
Systolic blood pressure | 3 months & 12 months
  Measured using an automated blood pressure monitor (in mm Hg)
Diastolic blood pressure | 3 months & 12 months
  Measured using an automated blood pressure monitor (in mm Hg)
Body mass index | 3 months & 12 months
  Calculated from weight (digital weight scale) and height (portable stadiometer) (in kg/m2)
Waist circumference | 3 months & 12 months
  Measured using tape measure (in cm)
Glycated hemoglobin (A1c) | 3 months & 12 months
  Measured using a point-of-care analyzer (%)
Daily steps | 3 months & 12 months
  Measured using a waist-worn accelerometer-based step counter over 7 days (average steps/day)
Total physical activity MET-minutes/week | 3 months & 12 months
  Measured using the International Physical Activity Questionnaire (IPAQ) - Short Form (sum of Walking + Moderate + Vigorous MET-minutes/week)
Vigorous physical activity MET-minutes/week | 3 months & 12 months
  Measured using the International Physical Activity Questionnaire (IPAQ) - Short Form (calculated as 8.0 * vigorous-intensity activity minutes * vigorous-intensity days)
Moderate physical activity MET-minutes/week | 3 months & 12 months
  Measured using the International Physical Activity Questionnaire (IPAQ) - Short Form (calculated as 4.0 * moderate-intensity activity minutes * moderate-intensity days)
Walking MET-minutes/week | 3 months & 12 months
  Measured using the International Physical Activity Questionnaire (IPAQ) - Short Version (calculated as 3.3 * walking minutes * walking days)
Total time spent sitting (on a week day) | 3 months & 12 months
  Measured using the Marshall Questionnaire (in minutes)
Healthful eating score | 3 months & 12 months
  Measured using the Starting the Conversation (STC) Questionnaire (summary score of 8 items; score range, 0-16; lower score indicates more healthful eating)
Fruit and vegetable intake | 3 months & 12 months
  Measured using the Canadian Community Health Survey
Sweetened sugary beverages intake | 3 months & 12 months
  Measured using the Behavioral Risk Factor Surveillance System Questionnaire
Total alcohol intake (weekly) | 3 months & 12 months
  Measured using a 7-day recall diary
Smoking status | 3 months & 12 months
  Measured using questions adapted from the Canadian Community Health Survey
Overall self-rated health status | 3 months & 12 months
  Measured using the EQ-5D 5 level version, specifically using the EQ visual analogue scale (EQ-VAS; range, 0-100; higher score indicates better self-rated health where 100 = best imaginable health state)
Well-being score | 3 months & 12 months
  Measured using the World Health Organization (Five) Well-Being Index (raw score is calculated from totalling 5 items and is converted to a percentage score when multiplied by 4; percentage score range, 0-100; higher score indicates better better quality of life where 100 represents best possible quality of life)
Social connectedness score | 3 months & 12 months
  Measured using the Duke Social Support Index (total score range, 11-33; higher values indicate higher levels of support)
Sleep quality global score | 3 months & 12 months
  Measured using the Pittsburgh Sleep Quality Index (calculated by totalling the sum of 7 component scores; score range, 0-21; higher scores indicate worse sleep quality)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Petrella, MD, PhD, Principal Investigator — Western University
Locations (40):
- United States (3):
  - Dort Federal Credit Union Event Center, Flint, Michigan
  - Saginaw Valley State University, Saginaw, Michigan
  - Veterans Memorial Coliseum, Portland, Oregon
- Canada (37):
  - City of Brooks, Brooks, Alberta
  - Mount Royal University, Calgary, Alberta
  - University of Lethbridge, Lethbridge, Alberta
  - Downtown Medicine Hat YMCA, Medicine Hat, Alberta
  - Northside Community Centre YMCA of Northern Alberta, Red Deer, Alberta
  - Club XO Fitness, Chilliwack, British Columbia
  - YMCA Kamloops, Kamloops, British Columbia
  - YMCA Okanagan, Kelowna, British Columbia
  - YMCA-YWCA Westhills, Langford, British Columbia
  - Langley Events Centre, Langley, British Columbia
  - Penticton Community Centre, Penticton, British Columbia
  - YMCA of Northern BC, Prince George, British Columbia
  - Shaw Centre, Salmon Arm, British Columbia
  - Avenir Centre, Moncton, New Brunswick
  - Afterburn Performance, Saint John, New Brunswick
  - YMCA of Halifax and Dartmouth, Halifax, Nova Scotia
  - Barrie YMCA, Barrie, Ontario
  - YMCA of Central Eastern Ontario - Belleville Branch, Belleville, Ontario
  - YMCA Sudbury, Greater Sudbury, Ontario
  - Les Chater Family YMCA, Hamilton, Ontario
  - YMCA of Kingston, Kingston, Ontario
  - A.R. Kaufman Family YMCA, Kitchener, Ontario
  - Bostwick YMCA, London, Ontario
  - Mississauga Burnhamthorpe Rd. YMCA Centre, Mississauga, Ontario
  - YMCA of North Bay, North Bay, Ontario
  - Oshawa Mary Street YMCA Centre, Oshawa, Ontario
  - YMCA of Owen Sound Grey Bruce, Owen Sound, Ontario
  - Balsillie Family YMCA, Peterborough, Ontario
  - YMCA Jerry McCaw Family Centre, Sarnia, Ontario
  - YMCA of Sault Ste Marie, Sault Ste. Marie, Ontario
  - Walker Family YMCA, St. Catharines, Ontario
  - YMCA at Central Park Athletics, Windsor, Ontario
  - University of Prince Edward Island, Charlottetown, Prince Edward Island
  - CBI Health Centre, Prince Albert, Saskatchewan
  - University of Regina, Regina, Saskatchewan
  - YMCA of Saskatoon, Saskatoon, Saskatchewan
  - Lt. Colonel Clifton Centre, Swift Current, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blunt WM, Kfrerer ML, Gill DP, Shillington KJ, Riggin B, Irwin JD, Bliss B, Petrella RJ. Process evaluation of the Hockey Fans in Training lifestyle intervention (for men with overweight or obesity). Transl Behav Med. 2025 Jan 16;15(1):ibaf002. doi: 10.1093/tbm/ibaf002. PMID 39963751
- [Derived] Petrella RJ, Gill DP, Boa Sorte Silva NC, Riggin B, Blunt WM, Kfrerer M, Majoni M, Marsh J, Irwin JD, Stranges S, Zwarenstein M, Zou G. The hockey fans in training intervention for men with overweight or obesity: a pragmatic cluster randomised trial. EClinicalMedicine. 2024 Nov 7;77:102911. doi: 10.1016/j.eclinm.2024.102911. eCollection 2024 Nov. PMID 39568632
- [Derived] Petrella RJ, Gill DP, Kfrerer M, Riggin B, Majoni M, Blunt W, Bliss B, Silva NCBS, Aspinall PS, Adekoya P, DiNunzio M, Marsh J, Zou G, Irwin JD. Hockey Fans in Training (Hockey FIT): Rationale, design, and baseline characteristics from a cluster randomized controlled trial in men with overweight or obesity. Contemp Clin Trials. 2023 Jun;129:107178. doi: 10.1016/j.cct.2023.107178. Epub 2023 Apr 7. PMID 37031793